CLINICAL TRIAL: NCT03837951
Title: Comparison of Figure-of-Eight Hand Measurements to Standard Volumetric Measurements and Its Reliability Within a Clinical Setting With Hand Injured Patients
Brief Title: Figure-of-Eight Hand, Volumetric Measurements and Reliability in Clinic With Hand Injured Patients
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Lowell (Other)
Responsible Party: Principal Investigator, ELewis, Associate Professor, Interim DPT Program Director, University of Massachusetts, Lowell
Other Study IDs: 11-056-LEW-XPD
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Hand Injuries; Edema Arm
Keywords: reliability; edema; physical therapy; occupational therapy; figure-of-eight
MeSH Terms: conditions — Hand Injuries; Edema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Uninjured hands: healthy participants without injuries to hands or wrists
  Interventions: Other: Figure-of-eight tape measure measurements on both hands; Other: Volumeter measurements
- Injured hands: participants undergoing medical treatment for recent hand or wrist injury
  Interventions: Other: Figure-of-eight tape measure measurements on both hands

INTERVENTIONS:
Other: Figure-of-eight tape measure measurements on both hands — Tape measure is wrapped around the wrist and hand and a measurement reading is taken. this is repeated 3 times.
Other: Volumeter measurements — Volumeter measurements to uninjured participants had 3 measurements taken of each hand.
  Groups: Uninjured hands

SUMMARY:
This study determined the intra-rater and inter-rater reliability of the Figure-of-Eight method on healthy hands, and compared the figure-of-eight measurements to the gold standard volumetric measurements. Part B of the study conducted in a clinic, assessed the intra-rater reliability and inter-rater reliability on both hands of patients with hand injuries.

DETAILED DESCRIPTION:
Edema is the retention of fluid in the intracellular spaces, which is common in inflammatory condition such as traumatic injury and post surgical conditions. Edema in the hand and wrist can result in detrimental physiological changes which decrease the range of motion of joint and limit the overall functional capacity and dexterity of the hand. The gold standard Volumetric measurements are reliable for measuring edema changes in upper extremity. Using volumeters can be cumbersome in a busy clinic. Figure-of-eight measurements using a tape measure on the wrist and hand is an easy way to measure edema and can capture the accumulation in the dorsal hand that circumferential tape measurements do not capture. This study was performed in two parts. Part A determined the intra-rater and inter-rater reliability of the Figure-of-Eight method on healthy hands, and compared the figure-of-eight measurements to the gold standard volumetric measurements. No study other study has compared right and left hands. Part B of the study was conducted in a clinic to assess the intra-rater reliability and inter-rater reliability on both hands of patients with hand injuries.

ELIGIBILITY:
Inclusion Criteria

* Healthy-part A
* Recent history of hand or wrist injury with swelling -part B

Exclusion Criteria

* Open wounds-part A
* Current swelling-part A
* History of injury in either upper extremity-part A
* Diabetes mellitus-part A
* Raynaud's Syndrome-part A
* Pregnant women-part A & B
* Could not speak English-part A & B
* Could not consent for oneself-part A & B

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Part A: Thirty healthy participants (10 men and 20 women) were recruited from the student population at a university.
  Part B: 17 participants with upper extremity injury (4 men & 13 women)
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2011-04-28 (Actual); Primary Completion 2014-04-30 (Actual); Study Completion 2014-04-30 (Actual)

PRIMARY OUTCOMES:
Figure-of-Eight non-injured hands | 1 day
  3 measurements of right and left hands of each non-injured participant by 3 hand therapists
Volumetric measurements on non-injured hands | 1 day
  3 measurements of right and left hands of each non-injured participant
Figure-of-Eight injured hands | 1 day
  3 measurements of right and left hands of each non-injured participant by 3 different hand therapists

CONTACTS AND LOCATIONS:
Overall Officials: Erika S. LEWIS, Ed.D, Principal Investigator — Associate Professor, University of Massachusetts Lowell

IPD SHARING:
Plan to Share IPD: No
Not planning to share the de-identified data on this population